CLINICAL TRIAL: NCT06844266
Title: Study on the Accuracy of the Association Between the "Physical Activity-Rating" and "Asthma Control Test" Questionnaires in the Anamnestic Evaluation of Asthma Symptom Control in Pediatric Patients
Brief Title: Accuracy of the Association Between the "PA-R" and "ACT" Questionnaires in Asthmatic Pediatric Patients
Acronym: QAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 7190
Record Dates: First submitted 2025-02-14; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Asthma in Children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma Control Test (ACT) + PA-R (Experimental): Association of "ACT + PA-R" questionnaires
  Interventions: Procedure: Administration of the ACT + PA-R questionnaires
- Asthma Control Test (ACT) (Active Comparator): ACT questionnaire
  Interventions: Procedure: ACT questionnaire

INTERVENTIONS:
Procedure: Administration of the ACT + PA-R questionnaires — The "ACT + PA-R" questionnaires will be administered to pediatric patients with a previously confirmed diagnosis of asthma, who attend the Pediatric Allergy Day Hospital for a routine check-up with spirometry before and after physical exertion.
  Arms: Asthma Control Test (ACT) + PA-R
Procedure: ACT questionnaire — The "ACT" questionnaire will be administered to pediatric patients with a previously confirmed diagnosis of asthma, who attend the Pediatric Allergy Day Hospital for a routine check-up with spirometry before and after physical exertion.
  Arms: Asthma Control Test (ACT)

SUMMARY:
A patient with asthma requires daily and long-term pharmacological treatment when symptoms are frequent and/or severe. International guidelines suggest increasing or reducing pharmacological therapy based on the individual's needs. On average, follow-up visits for a child with asthma treated with maintenance pharmacological therapy should be every 3 months. This period is often challenging to meet in clinical practice because of long waiting lists. An alternative solution could involve the use of structured questionnaires that the patient should fill out on their own (if aged 12 or older) or with the help of parents (if younger than 12). A similar solution is also suggested by international asthma guidelines. The doctor, upon receiving the questionnaire, for example through email, could make the appropriate management decisions and communicate them to the patient, again through email. For remote use, the test should have optimal sensitivity and specificity, otherwise, there is a risk of either underestimating or overestimating the need for adjustments to the maintenance therapy. The most commonly used is the Asthma Control Test (ACT), which did non demonstrate an elevated sensibility and specificity as revealed by different studies. Tripoli et al., for example, reported that 22% of children aged 12 or older with an ACT score = 25 have asthma and a fall in FEV1 >12% after physical exertion. Considering the information above, we considered combining the ACT with the Physical Activity-Rating (PA-R), a validated questionnaire for measuring the level of physical activity. It is possible that one of the issues lies in the lack of quantification of the patient's physical activity level when administering the ACT. Through an interventional study, our intention is to assess the diagnostic accuracy of the ACT + PA-R combination (test under experimentation) compared to ACT (traditional test) and compared to reference standard (spirometry before and after exertion). The goal of the study is to evaluate whether the combination of a high score in both the PA-R (>7) and ACT (>21) can accurately identify patients with well-controlled asthma, i.e., those with normal spirometry after physical exertion.

ELIGIBILITY:
Inclusion Criteria:

* Correctly diagnosed asthma;
* Age between 6 and 15 years;
* Understanding and signing of the informed consent by the parent/guardian;
* Understanding and signing of the assent by the minor.

Exclusion Criteria:

* Inability to correctly perform spirometry;
* Inability to correctly perform the exercise test;
* Unwillingness to sign the informed consent by the parent/guardian;
* Unwillingness to sign the assent by the minor.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the reliability of the single ACT test versus the combined test (ACT + PA-R) | 24 months
  One group of patients will be dministered the ACT test and one group the ACT + PAR test to compare the reliability between the two test and the reference standard (spirometry before and after physical exertion).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Miceli Sopo, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS